CLINICAL TRIAL: NCT05033704
Title: Effect of Human Plasma Protein Transfusion With and Without Crystalloids on Acid Base, Electrolytes and Tissue Perfusion During Major Liver Resection Surgeries
Brief Title: Effect of Human Plasma Protein Transfusion With and Without Crystalloids During Major Liver Resection Surgeries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MRC-01-18-256
Record Dates: First submitted 2021-07-28; First posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-07

CONDITIONS: Coagulation; Intravascular; Fluid Electrolyte Disorders
Keywords: Human Plasma Protein; Crystalloids; Liver Resection Surgeries
MeSH Terms: conditions — Thrombosis | interventions — plasma protein fraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (Group A) (Experimental): Twenty-four of the 48 patients will receive an intraoperative intravenous infusion of 5% human plasma protein fraction PPF, (A group). PPF 5% "Octapharma 5 %" is a colloid solution containing (47.6-52.5% proteins, of which 45.6-52.5 gm/L albumin and 142.5-157.5 mmol/L sodium).
  Fluids will be given targeting euvolemic state which is defined as central venous pressure (CVP) 5-10 mmHg or Stroke volume variation (SVV) of ≤ 13%. Central venous pressure (CVP) CVP of -1 to 1 mmHg or Stroke volume variation (SVV) of 18-21% (12) will be targeted during transaction times. The transfusion trigger will be Hemoglobin of ≤8 gm/dl.
  Interventions: Drug: 5% human plasma protein fraction (PPF)
- (Group RS) (No Intervention): 24 patients will receive an intraoperative intravenous infusion of crystalloids (0.9 % normal saline and/ or Lactated Ringer's solution) (RS group). Fluids will be given targeting euvolemic state which is defined as central venous pressure (CVP) 5-10 mmHg or Stroke volume variation (SVV) of ≤ 13%. Central venous pressure (CVP) CVP of -1 to 1 mmHg or Stroke volume variation (SVV) of 18-21% (12) will be targeted during transaction times. The transfusion trigger will be Hemoglobin of ≤8 gm/dl.

INTERVENTIONS:
Drug: 5% human plasma protein fraction (PPF) — Infusion of 5% human plasma protein fraction PPF. PPF 5% "Octapharma 5 %" is a colloid solution containing (47.6-52.5% proteins, of which 45.6-52.5 gm/L albumin and 142.5-157.5 mmol/L sodium).
  Other Names: 5% Human Albumen
  Arms: (Group A)

SUMMARY:
Evaluation of acid-base and electrolyte changes after administration of commonly used colloid solutions (plasma protein fraction contains 5% albumin), and crystalloids (saline 0.9% and lactated ringers solutions) is the primary endpoint of this study. The secondary endpoints are to study dilution acidosis and changes in plasma volume induced by albumin versus crystalloids and their effect on tissue perfusion by randomizing patients into two groups where each group receives intraoperatively one type of the two fluids. Changes in acid-base, electrolytes, and dilution acidosis

DETAILED DESCRIPTION:
To compare Between PPF 5% and crystalloids in the management of patients undergoing Liver resection and to conclude if any the benefits of treating those patients with high protein content fluids.

Methodology: Each patient will complete a full medical and surgical history and clinical examination.

Routine examinations will include complete blood picture, kidney function tests (serum urea, creatinine, sodium, and potassium), liver function tests (alanine transaminase, aspartate transaminase, prothrombin time and concentration and international normalized ratio, and serum albumin), random blood sugar, and serum electrolytes (Calcium, Chloride bicarbonate and lactate). Patients will be distributed randomly between two groups using a predetermined computer-generated randomized schedule. Twenty-four of the 48 patients will receive an intraoperative intravenous infusion of 5% human plasma protein fraction PPF, (A group). PPF 5%?Octapharma 5 %? is a colloid solution containing (47.6-52.5% proteins, of which 45.6-52.5 gm/L albumin and 142.5-157.5 mmol/L sodium). The remaining 24 patients will receive an intraoperative intravenous infusion of crystalloids (0.9 % normal saline and/ or Lactated Ringer's solution) (RS group). Fluids will be given targeting euvolemic state which is defined as central venous pressure (CVP) 5-10 mmHg or Stroke volume variation (SVV) of? 13%. Central venous pressure (CVP) CVP of -1 to 1 mmHg or Stroke volume variation (SVV) of 18-21% (12) will be targeted during transaction times.

The transfusion trigger will be Hemoglobin of? 8 gm/dl. Any patient who received additional blood products will be excluded from the study. General anesthesia will be induced using Propofol 2% and fentanyl. The ultrasound-guided central venous catheter will be inserted after induction of anesthesia in the right internal jugular vein. Arterial Cather size 20-gauge will be inserted in the radial artery. All patients will receive inhalational anesthesia using Sevoflurane, targeting MAC 1, and be ventilated using the Drager Xeus machine. Tidal volume of 7ml/Kg and zero PEEP will be used for all patients. All patients will receive furosemide 20-40 mg to maintain good diuresis and control central venous pressure. In addition to this, a 30-45 degree head-up position will be maintained. Arterial blood will be drawn through the radial artery catheter before the start of surgery and fluid infusion (time 0), the start of liver resection (time R), after Liver resection (time AR), and at the end of the procedure (time E). Arterial blood gas parameters (using atrial blood gas analyzer machine) including, pH, K+, Cl-, HCO3-, base deficit, and lactate concentrations will be measured. Hemoglobin, hematocrit concentrations, and albumin will be measured and recorded at time 0, R, AR & E. Intravascular albumin mass will be calculated based on plasma volume (PV) which will be calculated according to Nadler's Formula for calculating total blood volume in adult (TBV) (9, 14): PV = TBV ? (1 ? hematocrit)

ELIGIBILITY:
Inclusion Criteria:

* 18- 70 years old
* Not allergic to PPF5%, NS and RL,
* No morphological or functional cardiac valve/s changes, cardiac ischemia, significant arrhythmias or in failure,
* Patients with normal liver function tests before surgery and has no chronic active liver disease,
* Patients with normal kidney functions.

Exclusion Criteria:

* Patients with cardiac disease,
* Kidney disease,
* Liver dysfunction,
* Those who receive additional blood products other than PRBCs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2019-09-09 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Base deficit | Intra-operative at the end of the four stages of liver resection
  The primary end point of the study will be changes in base deficit in the two groups
Strong Ion difference | Intra-operative time at the end of four stages of liver resection
  The primary end point of the study will be changes in strong ion difference in the two groups
Intra-vascular Albumin content | Intra-operative time at the end of the four stages of liver resection
  The primary end point of the study will be changes in intra-vascular albumin mass in the two groups

SECONDARY OUTCOMES:
Kidney functions | Urine out put at the end of surgery and postoperative day one serum creatinine
  Two group comparison on postoperative serum creatinine and urine output at the end of surgery
Total blood loss | End of surgery blood loss
  Comparing the two groups regarding intra-operative blood loss
Changes in coagulation using Thromboelastogram | At the the end of resection phase and end of surgery
  Comparing the coagulation of the two groups at the end of resection and end of surgery
Tissue perfusion index | The four intra-operative stages of liver resection
  statistically comparing tissue perfusion index between the two groups at the 4 surgical times

CONTACTS AND LOCATIONS:
Overall Officials: Yasser Hammad, M.D., Principal Investigator — Hamad Medical Corporation - HMC
Locations (1):
- Hamad Medical Corporation, Doha, Baladīyat ad Dawḩah, Qatar

IPD SHARING:
Plan to Share IPD: Yes
A decision regarding sharing information will be taken at later stage
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Directly after IRB approval.
Access Criteria: Website

REFERENCES:
- [Background] Janeway, C. A.
- [Background] Greasley L, Russell RJ. Albumin and its role in trauma resuscitation. J R Army Med Corps. 2005 Jun;151(2):65-8. doi: 10.1136/jramc-151-02-01. No abstract available. PMID 16097108
- [Background] Ashraf S. Hasanin, Fatma M.A. Mahmoud, Hossam M. Soliman. Factors affecting acid base status during hepatectomy in cirrhotic patients. Egyptian Journal of Anesthesia (2013) 29, 305-310).
- [Result] Semin Thromb Hemost 1980; 6(2): 85-120 DOI: 10.1055/s-2007-1005097
- [Result] Peters T Jr. Serum albumin. Adv Protein Chem. 1985;37:161-245. doi: 10.1016/s0065-3233(08)60065-0. No abstract available. PMID 3904348
- [Result] Quinlan GJ, Martin GS, Evans TW. Albumin: biochemical properties and therapeutic potential. Hepatology. 2005 Jun;41(6):1211-9. doi: 10.1002/hep.20720. No abstract available. PMID 15915465
- [Result] Tullis JL. Albumin. 1. Background and use. JAMA. 1977 Jan 24;237(4):355-60 CONTD. doi: 10.1001/jama.237.4.355. No abstract available. PMID 576167
- [Result] Liumbruno GM, Bennardello F, Lattanzio A, Piccoli P, Rossettias G; Italian Society of Transfusion Medicine and Immunohaematology (SIMTI). Recommendations for the use of albumin and immunoglobulins. Blood Transfus. 2009 Jul;7(3):216-34. doi: 10.2450/2009.0094-09. No abstract available. PMID 19657486
- [Result] Pusey C, Dash C, Garrett M, Gascoigne E, Gesinde M, Gillanders K, Wallington T. Experience of using human albumin solution 4.5% in 1195 therapeutic plasma exchange procedures. Transfus Med. 2010 Aug 1;20(4):244-9. doi: 10.1111/j.1365-3148.2010.00999.x. Epub 2010 Mar 11. PMID 20230532
- [Result] Dill DB, Costill DL. Calculation of percentage changes in volumes of blood, plasma, and red cells in dehydration. J Appl Physiol. 1974 Aug;37(2):247-8. doi: 10.1152/jappl.1974.37.2.247. No abstract available. PMID 4850854
- [Result] Goodkin DA, Raja RM, Saven A. Dilutional acidosis. South Med J. 1990 Mar;83(3):354-5. doi: 10.1097/00007611-199003000-00029. PMID 2315790
- [Result] Mathes DD, Morell RC, Rohr MS. Dilutional acidosis: is it a real clinical entity? Anesthesiology. 1997 Feb;86(2):501-3. doi: 10.1097/00000542-199702000-00028. No abstract available. PMID 9054271
- [Result] Dunki-Jacobs EM, Philips P, Scoggins CR, McMasters KM, Martin RC 2nd. Stroke volume variation in hepatic resection: a replacement for standard central venous pressure monitoring. Ann Surg Oncol. 2014 Feb;21(2):473-8. doi: 10.1245/s10434-013-3323-9. Epub 2013 Oct 23. PMID 24150192
- [Result] Norberg A, Rooyackers O, Segersvard R, Wernerman J. Leakage of albumin in major abdominal surgery. Crit Care. 2016 Apr 26;20(1):113. doi: 10.1186/s13054-016-1283-8. PMID 27117323
- [Result] Nadler SB, Hidalgo JH, Bloch T. Prediction of blood volume in normal human adults. Surgery. 1962 Feb;51(2):224-32. No abstract available. PMID 21936146